CLINICAL TRIAL: NCT03234699
Title: The Effect of Multiple Doses of Cenobamate (YKP3089) on the Single Dose Pharmacokinetics of Cytochrome P450 Substrates (midazolam, Warfarin, Omeprazole and Bupropion) Administered Orally in an Open-label, One-sequence Study in Healthy Subjects
Brief Title: Assess the Influence of Cenobamate on the PK of Cytochrome P450 (CYP) Probe Drugs As a Means of Predicting Drug-drug Interactions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YKP3089C026
Record Dates: First submitted 2017-04-17; First posted 2017-07-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — Cenobamate; Midazolam; Warfarin; Omeprazole; Bupropion

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Group (Experimental)
  Interventions: Drug: Cenobamate; Drug: midazolam; Drug: Warfarin Pill; Drug: Omeprazole Pill; Drug: Bupropion Pill

INTERVENTIONS:
Drug: Cenobamate — 12.5 mg q.d.(Days 13-26), 25 mg q.d. (Days 27-40), 50 mg q.d. (Days 41-54), 100 mg q.d. (Days 55-70), 150 mg q.d. (Days 71-84), 200 mg q.d. (Days 85-110)
Drug: midazolam — 2 mg midazolam syrup (Days 7, 69, 105)
Drug: Warfarin Pill — 5 mg (Days 7 and 105)
Drug: Omeprazole Pill — 20 mg (Days 7 and 105)
Drug: Bupropion Pill — 150 mg (Days 1 and 99)

SUMMARY:
This study is aimed to investigate the influence of cenobamate on the activity of CYP3A4/5, CYP2B6, CYP2C19, and CYP2C9 by using drugs recommended by both the FDA and EMA as in vivo probes. In order to avoid a potential pharmacokinetic interaction between the probes, midazolam (CYP3A), warfarin (CYP2C9), and omeprazole (CYP2C19) will be administered together as a validated cocktail and separately from bupropion (CYP2B6) using an adequate washout time period between the 2 assessments.

The starting daily dose of cenobamate will be 12.5 mg, which will be administered for 2 weeks. Then, daily cenobamate doses will be increased every 2 weeks to 25 mg, 50 mg, 100 mg, 150 mg, and 200 mg. The CYP probes will be tested before cenobamate administration, at steady state at 100mg/day of cenobamate for midazolam only and finally at steady state at 200mg/day of cenobamate for all CYP probes.

The results of this DDI study will provide a basis to make appropriate dose recommendation for a safe use of concomitant drugs with cenobamate using these isoenzymes in their metabolic pathway.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 to 50 years of age inclusive
2. Subject is willing and able to provide informed consent
3. Body mass index (BMI) within 19.0 kg/m2 and 29.9 kg/m2, inclusive, at screening
4. Subject is a non- or ex-smoker and has not used any nicotine containing products within 6 months prior to screening
5. Subjects who are considered generally healthy upon completion of medical history, physical examination, vital signs, screening laboratory results and screening ECG in the opinion of the Investigator
6. Subjects who are willing and able to comply with the dosing/visit schedule, laboratory tests, pharmacokinetic sampling schedule, and other study procedures
7. A female study subject must meet one of the following criteria:

   If of childbearing potential - agrees to use one of the accepted contraceptive regimens from screening, during the study and for at least 30 days after the last dose of the study medication. Hormonal contraceptives alone will not be considered an adequate method of contraception. An acceptable method of contraception includes one of the following:
   1. Diaphragm and spermicide
   2. Condom with spermicide
   3. Sponge and spermicide
   4. Intrauterine device (with or without hormones; placement at least 3 months prior to Screening) in combination with a barrier method
   5. Oral contraceptives, Depo-Provera, Norplant, Patch or intrauterine progesterone contraceptive for at least 90 days prior to screening in combination with a barrier method.
   6. Vasectomized partner (6 months minimum since vasectomy)
   7. Complete abstinence from heterosexual intercourse. However, if the subject becomes sexually active, 1 of the above methods must be utilized.

   If a female of non-childbearing potential - should be surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation at least 6 months prior to Screening) or in a menopausal state (at least 1 year without menses), as confirmed by FSH levels (post menopausal must be confirmed by the subject having a serum follicle stimulating hormone greater than 40mIU/ml at screening)
8. A female study subject must agree not to donate eggs during the study and for at least 30 days after the last dose of the study medication
9. A male study subject must agree to use one of the accepted contraceptive regimens during the study and for at least 90 days after the last dose of the study medications;

   1. Abstinence from heterosexual intercourse. However, if the subject becomes sexually active, 1 of the below methods must be utilized
   2. Female partner with hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch) in combination with a barrier method
   3. Female partner with intrauterine device (with or without hormones) in combination with a barrier method
   4. Female partner with condom with spermicide used by male study subject
   5. Female partner of non-childbearing potential
   6. Female partner with diaphragm with spermicide
   7. Female partner with sponge and spermicide
   8. Male sterilization with absence of sperm in the post vasectomy ejaculate for ≥ 6 months
10. A male study subject must agree not to donate sperm during the study and for at least 90 days after the last dose of the study medication

Exclusion Criteria:

1. Females who are breastfeeding
2. Inadequate venous access
3. History of any drug related hypersensitivity reactions as well as severe hypersensitivity reactions (like angioedema), or DRESS syndrome to any drugs in the opinion of the Investigator
4. History of 1st degree relative having a serious cutaneous adverse reaction
5. Current clinically significant rash
6. Clinically significant history or evidence of gastrointestinal, hepatic, renal, endocrine, pulmonary, neurological, psychiatric, cardiovascular, hematologic, dermatologic, immunologic disease or any other condition known to interfere with the absorption, distribution, metabolism or elimination of drugs that in the opinion of the Investigator would jeopardize the safety of the subject or impact validity of study results
7. History of hepatic impairment, cholecystectomy, renal impairment or any other condition known to interfere with the absorption, distribution, metabolism or elimination of orally administered drug
8. Presence of observed abnormality (evidenced from physical examination, ECG, vital signs, or laboratory evaluation) that would be clinically significant in the opinion of the Investigator
9. Current evidence or history of suicidal tendency, seizures, state of confusion or any other clinically relevant psychiatric disease.
10. Subject is at imminent risk of suicide (positive response to question 4 or 5 on the C-SSRS) or had a suicide attempt within 6 months prior to the screening visit
11. History of regular alcohol consumption exceeding 7 drinks per week for females and 14 drinks per week for males within 6 months prior to screening
12. Has current or recent history (within the past year) of alcohol or drug abuse or dependence
13. Any clinically significant illness in the previous 30 days prior to screening
14. Use of any enzyme-modifying drugs, including strong inhibitors of CYP enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem, and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort) in the previous 30 days prior to Day 1 of this study
15. Use of all drugs associated with DRESS syndrome such as phenobarbital, carbamazepine, phenytoin, lamotrigine, minocycline, sulfonamides, allopurinol, modafinil, dapsone, ziprasidone, vancomycin and olanzapine in the previous 6 months prior to Day 1 of this study
16. Clinically-relevant, unusual dietary habits (e.g., vegan, Atkins), dietary restrictions, and/or food allergies
17. Positive urine screen for alcohol and/or drugs of abuse at screening and at each admission
18. Positive test results for HIV-1/HIV-2 Antibodies, Hepatitis B surface Antigen (HBsAg) or Hepatitis C Antibody (HCVAb) at screening
19. Has been administered any investigational drug 30 days (or 6 times its terminal half-live) prior to Day 1 of this study
20. Females with a positive pregnancy test at screening, regardless of child-bearing potential prior to Day 1 of this study
21. Blood donation (excluding plasma donation) of approximately 500 mL within 56 days prior to screening
22. Subject is unlikely to comply with the study protocol or, in the opinion of the Investigator, would not be a suitable candidate for participation in the trial
23. Anyone who has previously been exposed to cenobamate (prior to participation in this study)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters AUC | bupropion (6 days), midazolam (24 hrs), omeprazole (24 hrs), warfarin (7 days)
  Will be determined for S- and R-bupropion, total bupropion, midazolam, S-warfarin and R-warfarin, and omeprazole when administered with and without cenobamate at steady state
Pharmacokinetic parameters Cmax | bupropion (6 days), midazolam (24 hrs), omeprazole (24 hrs), warfarin (7 days)
  Will be determined for S- and R-bupropion, total bupropion, midazolam, S-warfarin and R-warfarin, and omeprazole when administered with and without cenobamate at steady state

SECONDARY OUTCOMES:
Pharmacokinetic parameters AUC | bupropion (6 days), midazolam (24 hrs), omeprazole (24 hrs), warfarin (7 days)
  Will be determined for probe drug metabolites (S,S-hydroxybupropion and R,R-hydroxybupropion, threohydrobupropion, 1-hydroxymidazolam, and 5-OH omeprazole)
Pharmacokinetic parameters Cmax | bupropion (6 days), midazolam (24 hrs), omeprazole (24 hrs), warfarin (7 days)
  Will be determined for probe drug metabolites (S,S-hydroxybupropion and R,R-hydroxybupropion, threohydrobupropion, 1-hydroxymidazolam, and 5-OH omeprazole)
Pharmacokinetic parameters AUC (to infinity) | bupropion (6 days), midazolam (24 hrs), omeprazole (24 hrs), warfarin (7 days)
  Will be determined for probe drug metabolites (S,S-hydroxybupropion and R,R-hydroxybupropion, threohydrobupropion, 1-hydroxymidazolam, and 5-OH omeprazole)
Pharmacokinetic parameter RAUC (ratio of metabolite to parent) | bupropion (6 days), midazolam (24 hrs), omeprazole (24 hrs), warfarin (7 days)
  Will be determined for 5-OH omeprazole/omeprazole, 1-OH midazolam/midazolam, S,S-OH-bupropion/S-bupropion, R,R-OH-bupropion/R-bupropion, total OH-bupropion/total bupropion, threohydrobupropion/R-bupropion

OTHER OUTCOMES:
Pharmacokinetic parameters tmax | bupropion (6 days), midazolam (24 hrs), omeprazole (24 hrs), warfarin (7 days)
  Will be determined for the probe drugs (and metabolites) when administered with or without cenobamate at steady state
Pharmacokinetic parameters Ctz | bupropion (6 days), midazolam (24 hrs), omeprazole (24 hrs), warfarin (7 days)
  Will be determined for the probe drugs (and metabolites) when administered with or without cenobamate at steady state
Pharmacokinetic parameters tz | bupropion (6 days), midazolam (24 hrs), omeprazole (24 hrs), warfarin (7 days)
  Will be determined for the probe drugs (and metabolites) when administered with or without cenobamate at steady state
Pharmacokinetic parameters t1/2 | bupropion (6 days), midazolam (24 hrs), omeprazole (24 hrs), warfarin (7 days)
  Will be determined for the probe drugs (and metabolites) when administered with or without cenobamate at steady state
Pharmacokinetic parameters CL/F | bupropion (6 days), midazolam (24 hrs), omeprazole (24 hrs), warfarin (7 days)
  Will be determined for the probe drugs (and metabolites) when administered with or without cenobamate at steady state
Pharmacokinetic parameters Vz/F | bupropion (6 days), midazolam (24 hrs), omeprazole (24 hrs), warfarin (7 days)
  Will be determined for the probe drugs (and metabolites) when administered with or without cenobamate at steady state
Pharmacokinetic parameters Cmin | bupropion (6 days), midazolam (24 hrs), omeprazole (24 hrs), warfarin (7 days)
  Will be determined for the probe drugs (and metabolites) when administered with or without cenobamate at steady state

CONTACTS AND LOCATIONS:
Locations (1):
- Vince and Associates Clinical Research, Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No